CLINICAL TRIAL: NCT06710275
Title: Étude rétrospective de la Valeur Pronostique du pCO2 Gap Durant la Circulation Extracorporelle en Chirurgie Cardiaque
Brief Title: Pronostic Value of Gap CO2 During Cardiac Pulmonary Bypass in Cardiac Surgery: a Multicenter Retrospective Study
Acronym: CO2-CARD
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP241392
Record Dates: First submitted 2024-11-08; First posted 2024-11-29 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Cardiac Surgery Associated Kidney Injury
Keywords: Cardiac surgery; AKI; Cardiopulmonary bypass

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- elevated gap CO2 group and low gap CO2 group: Gap CO2 is calculated as PvCO2-PaCO2, using arterial and venous blood gases taken during CPB. Patients will be included in the elevated gap CO2 group when gap CO2 during CPB is > 6 mmHg

SUMMARY:
Cardiac surgery associated acute kidney injury (CSA-AKI) is one of the most frequent and severe complications after cardiac surgery. The association between acute kidney injury and the mismatch between oxygen consumption and delivery has been well established during cardiopulmonary bypass (CPB) and contributes to the development of CSA-AKI. In this study, the investigators aim to explore the use of gap CO2 during cardiac surgery and its relation with CSA-AKI. In order to explore this association, the invetigators built a retrospective, multicentric study. All patient who underwent cardiac surgery with cardiopulmonary bypass in two French ICU between 03/2019 and 04/2023 and for which information about gap CO2 during CPB is available will be included. After inclusion, patient will be divided in two groups according to the presence or absence of an elevated gap CO2. Occurence of CSA-AKI and other outcomes will be compared between groups, using multivariate analysis.

DETAILED DESCRIPTION:
Cardiac surgery associated acute kidney injury (CSA-AKI) is one of the most frequent and severe complications after cardiac surgery. The association between acute kidney injury and the mismatch between oxygen consumption and delivery has been well established during cardiopulmonary bypass (CPB) and contributes to the development of CSA-AKI. In order to explore this association, investigators build a retrospective study including all patients who underwent cardiac surgery requiring CPB in two French hospitals and for which data about gap CO2 during CPB is available. Patients will be divided into two groups according to the presence or absence of an elevated gap CO2 during CPB, defined as > 6 mmHg. The primary outcome is the occurrence of CSA-AKI, defined by KDIGO recommendations, according gap CO2. Secondary outcomes include others post-operative complications as defined by international guidelines. Performance of gap CO2 to predict CSA-AKI will be evaluated by calculating the Area Under the Curve (AUC) of the associated ROC curve. We'll also assess the correlation between gap CO2 and other perfusion parameters (lactate, svO2) and with mean DO2 during CPB.

ELIGIBILITY:
Inclusion criteria:

1. Informed patients who did not object to the use of their data in the study.
2. Patients undergoing cardiac surgery with extracorporeal circulation.
3. Patients for whom a pCO2 gap measurement is available during ECG.

Non-inclusion criteria :

1. Heart transplant patients
2. Patients who have received long-term cardiac assistance
3. Minor patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients older than 18, which underwent cardiac surgery with cardiopulmonary bypass
Sampling Method: Non-Probability Sample
Enrollment: 318 (Actual)
Dates: Start 2025-02-27 (Actual); Primary Completion 2025-04-04 (Actual); Study Completion 2025-04-04 (Actual)

PRIMARY OUTCOMES:
Acute Kidney Injury | within the 7 days after surgery
  proportion of patient with acute kidney injury of Acute Kidney Injury as defined in the KDIGO guidelines within the first 7 days after the cardiac surgery

SECONDARY OUTCOMES:
Mortality, occurrence of other complications | within the 28 days after surgery
  proportion of patient with others post-operative complications as defined by international post-operative guidelines: atrial fibrillation, ARDS , VA-ECMO implantation, cardiac arrest, length of stay in ICU and hospital and the mortality rate within the first 28 days

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Service d'Anesthésie Réanimation, Hôpital de la Pitié-Salpêtrière, Paris
  - Service d'Anesthésie-Réanimation, Hôpital Pontchaillou, Rennes, Rennes

IPD SHARING:
Plan to Share IPD: Yes
The procedures carried out with the French data privacy authority (CNIL, Commission nationale de l'informatique et des libertés) do not provide for the transmission of the database, nor do the information and consent documents signed by the patients.
  Consultation by the editorial board or interested researchers of individual participant data that underlie the results reported in the article after deidentification may nevertheless be considered, subject to prior determination of the terms and conditions of such consultation and in respect for compliance with the applicable regulations.
Supporting Information: Study Protocol
Time Frame: Beginning 3 months and ending 3 years following article publication. Requests out of these time frame can also be submitted to the sponsor
Access Criteria: Researchers who provide a methodologically sound proposal.